CLINICAL TRIAL: NCT05156996
Title: A Prospective Real-World Multi-Center Post-Market Observational Evaluation of Supersaturated O2 Therapy Using the TherOx® Downstream® System After PCI vs. PCI Alone Among Patients Undergoing PCI for Acute Anterior Myocardial Infarction
Brief Title: A Prospective Real-World Multi-Center Post-Market Observational Evaluation of Supersaturated O2 Therapy Using the TherOx® Downstream® System
Acronym: REAL
Status: Terminated | Type: Observational
Why Stopped: Transitioning to a new Registry trial
Sponsor: TherOx (Industry)
Responsible Party: Sponsor
Other Study IDs: REAL SSO2
Record Dates: First submitted 2021-11-02; First posted 2021-12-14 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Anterior Acute Myocardial Infarction (AMI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Treatment Group
  Interventions: Device: Supersaturated O2 Therapy of the Therox Downstream System®
- Control Group
  Interventions: Procedure: PCI alone

INTERVENTIONS:
Device: Supersaturated O2 Therapy of the Therox Downstream System® — SuperSaturated Oxygen Therapy (SSO2 Therapy) to targeted ischemic regions perfused by the patient's left anterior descending coronary artery immediately following revascularization by means of percutaneous coronary intervention (PCI) with stenting that has been completed within 6 hours after the onset of anterior myocardial infarction (AMI) symptoms caused by a left anterior descending artery infarct lesion.
  Groups: Treatment Group
Procedure: PCI alone — Percutaneous Coronary Intervention for treatment of acute MI
  Groups: Control Group

SUMMARY:
The purpose of this study is to collect real-world data on the TherOx DownStream System® to assess the effectiveness and cost- effectiveness of SSO2 Therapy, compared with PCI alone for treatment of patients with acute anterior MI.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 years or older.
2. Presentation with anterior acute ST-elevation myocardial infarction (> 1 mm ST-segment elevation in two or more contiguous leads between V1 and V4).
3. The primary stented infarct-related lesion(s) must be in the proximal and/or mid-LAD coronary artery (other lesions may be treated if clinically indicated).
4. Successful angioplasty within 6 hours of symptom onset, as documented by <50% diameter residual angiographic stenosis within all treated culprit lesions with TIMI 2 or 3 flow and no major complications such as perforation or shock.
5. The patient or their legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided and signed written informed consent, approved by the appropriate Institutional Review Board (IRB).
6. Patient and his/her physician agree to all required follow-up procedures and visits.

Exclusion Criteria:

1. Ipsilateral insertion of a second sheath in a single femoral artery for SuperSaturated Oxygen Therapy is strictly contraindicated.
2. Presence of an intra-aortic balloon pump.
3. Proximal coronary stenosis that would restrict flow with the SSO2 Catheter in place
4. Presence of a post-intervention non-stented coronary dissection or perforation.
5. Cardiac valvular stenosis or insufficiency, pericardial disease or non-ischemic cardiomyopathy.
6. Pregnant or nursing women.
7. Cardiogenic shock.
8. Patients contraindicated for anticoagulation therapy.
9. Patients with ventricular pseudoaneurysm, VSD, or severe mitral valve regurgitation (with or without papillary muscle rupture).
10. Hemoglobin < 10 g/dL.
11. Gastrointestinal or genitourinary bleeding within the last two months, or any major surgery (including CABG) within six weeks of procedure.
12. Patients with active COVID-19 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who meets the protocol defined eligibility criteria and none of the exclusion criteria at the time of completion of index procedure and who consents to participate.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-12-04 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Measures (hierarchical) at 12-months post-procedure include rates of: | 12 months post-procedure
  Rate of Cardiovascular Death
Measures (hierarchical) at 12-months post-procedure include rates of: | 12 months post-procedure
  Rate of Heart Transplant or LVAD
Measures (hierarchical) at 12-months post-procedure include rates of: | 12 months post-procedure
  Rate of ICD/CRT device implanted
Measures (hierarchical) at 12-months post-procedure include rates of: | 12 months post-procedure
  Rate of Rehospitalization for heart failure between discharge and 12 months post-procedure
Measures (hierarchical) at 12-months post-procedure include rates of: | 12 months post-procedure
  Rate of KCCQ-OS score at 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Charleston Area Medical Center, Charleston, West Virginia
  - St. Mary's Medical Center, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided